CLINICAL TRIAL: NCT04517253
Title: A Phase 2/3, Multicenter, Open-Label Study to Evaluate the Efficacy and Safety of Baricitinib in Adult and Pediatric Japanese Patients With NNS/CANDLE, SAVI, and AGS
Brief Title: A Study of Baricitinib (LY3009104) in Adult and Pediatric Japanese Participants With NNS/CANDLE, SAVI, and AGS
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: The study was terminated due to efficacy/effectiveness reasons
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17571; I4V-JE-JAJE (Other: Eli Lilly and Company); 2025-000001-16 (EudraCT Number)
Record Dates: First submitted 2020-08-17; First posted 2020-08-18 (Actual); Results first posted 2022-12-21 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-06

CONDITIONS: Nakajo-Nishimura Syndrome; Chronic Atypical Neutrophilic Dermatosis With Lipodystrophy and Elevated Temperature Syndrome; STING-Associated Vasculopathy With Onset in Infancy; Aicardi Goutieres Syndrome
Keywords: Nakajo-Nishimura Syndrome; CANDLE; SAVI; AGS
MeSH Terms: conditions — Nakajo syndrome; Aicardi-Goutieres syndrome | interventions — baricitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- CANDLE (Experimental): Participants with chronic atypical neutrophilic dermatosis with lipodystrophy and elevated temperature (CANDLE) were administered an optimized final dosage of baricitinib, ranging from 8 mg to 12 mg daily (initially 8 mg, with gradual escalation to 10 mg and 12 mg), either as tablets or oral suspension, for 12 weeks. This dosage was determined during a prior 8-week dose-adjustment period, tailored to each participant's weight and estimated glomerular filtration rate (eGFR). Participants then continued receiving baricitinib at their optimized dosage for 191.1 weeks.
  Interventions: Drug: Baricitinib
- SAVI (Experimental): Participants with stimulator of interferon genes (STING)-associated vasculopathy with onset during infancy (SAVI) were administered an optimized final dosage of baricitinib, ranging from 6 mg to 12 mg daily (initially 6 mg, with gradual escalation to 8 mg, 10 mg, and 12 mg), either as tablets or oral suspension, for 24 weeks. This dosage was determined during a prior 8-week dose-adjustment period, tailored to each participant's weight and eGFR. Participants then continued receiving baricitinib at their optimized dosage for 202.9 weeks.
  Interventions: Drug: Baricitinib
- Aicardi-Goutières Syndrome (AGS) (Experimental): Participants with Aicardi-Goutières Syndrome (AGS) were administered an optimized final dosage of baricitinib, ranging from 6 mg to 8 mg daily (initially 6 mg, with gradual escalation to 8 mg), either as tablets or oral suspension, for 24 weeks. This dosage was determined during a prior 8-week dose-adjustment period, tailored to each participant's weight and eGFR. Participants then continued receiving baricitinib at their optimized dosage for 206.1 weeks.
  Interventions: Drug: Baricitinib

INTERVENTIONS:
Drug: Baricitinib — Administered orally
  Other Names: LY3009104

SUMMARY:
The main purpose of this study is to evaluate the efficacy and safety of baricitinib in adult and pediatric Japanese participants with Nakajo-Nishimura Syndrome/chronic atypical neutrophilic dermatosis with lipodystrophy and elevated temperature (NNS/CANDLE), STING-associated vasculopathy with onset during infancy (SAVI), and Aicardi-Goutières Syndrome (AGS).

ELIGIBILITY:
Inclusion Criteria:

* Have systemic signs and symptoms of inflammation as manifested NNS/CANDLE, SAVI, AGS
* Have been diagnosed with genetic diagnosis
* Men must agree to use a reliable method of birth control during the study
* Women not of child-bearing potential or nonbreastfeeding
* Women must agree to use birth control or remain abstinent during the study and for at least 12 weeks after stopping treatment
* NNS/CANDLE and SAVI patients who are ≥17.5 months of age
* AGS patients who are ≥6 months of age
* Are ≥ 5kg in body weight

Exclusion Criteria:

* Have received immunosuppressive biologic agent/monoclonal antibody/oral JAK inhibitor/OAT3 inhibitor and cannot discontinue prior to investigational product initiation. Note: A washout period is required to each drug.
* Have diagnosis of current active tuberculosis (TB) or, latent TB who did not receive appropriate treatment.
* Have had a serious infection within 12 weeks prior to screening.
* Have a history of lymphoproliferative disease
* Have any history of venous thromboembolic event (VTE) (deep vein thrombosis [DVT]/pulmonary embolism [PE]) prior to screening.
* Have had any major surgery within 8 weeks prior to screening.
* Have previously been enrolled in any other study investigating baricitinib.

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-10-27 (Actual); Primary Completion 2023-04-04 (Actual); Study Completion 2024-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (5):
- Japan (5):
  - Nara Medical University Hospital, Kashihara, Nara
  - Tokyo Medical And Dental University Medical Hospital, Bunkyō, Tokyo
  - National Center For Child Health And Development, Setagaya-ku, Tokyo
  - Hiroshima University Hospital, Hiroshima
  - Wakayama Medical University Hospital, Wakayama

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- [Derived] Kanazawa N, Ishii T, Takita Y, Nishikawa A, Nishikomori R. Efficacy and safety of baricitinib in Japanese patients with autoinflammatory type I interferonopathies (NNS/CANDLE, SAVI, And AGS). Pediatr Rheumatol Online J. 2023 Apr 22;21(1):38. doi: 10.1186/s12969-023-00817-8. PMID 37087470
- See also: A Study of Baricitinib (LY3009104) in Adult and Pediatric Japanese Participants With NNS/CANDLE, SAVI, and AGS — https://trials.lillytrialguide.com/en-US/trial/4deb45sM6OlbQ6MBzCAx6H

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Per analysis plan,only for participants with chronic atypical neutrophilic dermatosis with lipodystrophy and elevated temperature (CANDLE),a pretreatment period lasted for 12 weeks, during which natural history data were collected.This data serves as baseline to assess changes during baricitinib treatment for evaluating key secondary outcomes: Percentage of days with a mean daily symptom score below 0.5,Average daily symptom score,and the Physician's Global Assessment of Disease Activity scores.
Pre-assignment Details: Participants who met all eligibility criteria underwent an 8-week dose adjustment period and received an optimized dosage of baricitinib during the primary treatment period (12 weeks [week 8 to week 20] for CANDLE and 24 weeks [week 8 to week 32] for SAVI or AGS participants), followed by a maintenance period of up to 191.1 weeks for CANDLE participants, and up to 202.9 weeks for SAVI participants, and up to 206.1 weeks for AGS participants.
Period: Primary Treatment Period
Arm/Group | CANDLE | SAVI | Aicardi-Goutières Syndrome (AGS)
Started | 5 | 3 | 2
Received at Least One Dose of Study Drug | 5 | 3 | 2
Completed | 4 | 2 | 2
Not Completed | 1 | 1 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Death | 0 | 1 | 0
Period: Maintenance Period
Arm/Group | CANDLE | SAVI | Aicardi-Goutières Syndrome (AGS)
Started | 4 | 2 | 2
Completed | 0 | 0 | 0
Not Completed | 4 | 2 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Study Terminated by Sponsor | 3 | 2 | 2

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least one dose of study drug.
Groups:
- CANDLE: Participants with CANDLE were administered an optimized final dosage of baricitinib, ranging from 8 mg to 12 mg daily (initially 8 mg, with gradual escalation to 10 mg and 12 mg), either as tablets or oral suspension, for 12 weeks. This dosage was determined during a prior 8-week dose-adjustment period, tailored to each participant's weight and eGFR. Participants then continued receiving baricitinib at their optimized dosage for 191.1 weeks.
- SAVI: Participants with SAVI were administered an optimized final dosage of baricitinib, ranging from 6 mg to 12 mg daily (initially 6 mg, with gradual escalation to 8 mg, 10 mg, and 12 mg), either as tablets or oral suspension, for 24 weeks. This dosage was determined during a prior 8-week dose-adjustment period, tailored to each participant's weight and eGFR. Participants then continued receiving baricitinib at their optimized dosage for 202.9 weeks.
- Aicardi-Goutières Syndrome (AGS): Participants with AGS were administered an optimized final dosage of baricitinib, ranging from 6 mg to 8 mg daily (initially 6 mg, with gradual escalation to 8 mg), either as tablets or oral suspension, for 24 weeks. This dosage was determined during a prior 8-week dose-adjustment period, tailored to each participant's weight and eGFR. Participants then continued receiving baricitinib at their optimized dosage for 206.1 weeks.
- Total: Total of all reporting groups
Arm/Group | CANDLE | SAVI | Aicardi-Goutières Syndrome (AGS) | Total
Number analyzed (Participants) | 5 | 3 | 2 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.20 (13.79) | 9.70 (9.81) | 7.50 (2.12) | 24.00 (19.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 1 | 5
  Male | 4 | 0 | 1 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 3 | 2 | 10
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 5 | 3 | 2 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Japan | 5 | 3 | 2 | 10
Weight [Count of Participants; unit: Participants]
  >=10 -<20 | 0 | 2 | 2 | 4
  >=40 -<50 | 4 | 1 | 0 | 5
  >=50 -<60 | 1 | 0 | 0 | 1
Baseline estimated glomerular filtration rate (eGFR) [Mean (Standard Deviation); unit: mL/min/1.73m^2] — Due to character constraint unit of measure expanded here as milliliter per minute per 1.72 meter square (mL/min/1.73m^2)
  mL/min/1.73m^2 | 124.69 (19.32) | 109.37 (22.50) | 99.80 (9.77) | 115.11 (20.08)
Mean Daily Diary Score [Mean (Standard Deviation); unit: score on a scale] — Diaries were specific to conditions (NNS/CANDLE, SAVI, AGS). For NNS/CANDLE, participants rated symptoms (fever, rash, pain, headache, fatigue), and for SAVI, participants rated symptoms (fever, rash, pain, fatigue, respiratory issues, ulcers) on a scale from 0 (no symptoms) to 4 (severe). The mean daily score range was 0-4, with higher scores indicating more severe symptoms. For AGS, symptoms (neurologic disability, crying, sleep, seizures, fever, irritability, skin findings) were rated similarly. The mean daily score range was 0-4.25. Total score was not utilized. Population: The questionnaire in the daily diary score differs among diseases (CANDLE, SAVI, and AGS), and we cannot calculate a total score. Hence, data are reported separately, and 0 is entered for the Numbers Analyzed for the Arms/Groups to which a particular row does not apply for each Baseline Measure.
  score on a scale
    CANDLE: number analyzed (Participants) | 5 | 0 | 0 | 5
    CANDLE | 0.92 (0.345) |  |  | 0.92 (0.345)
    SAVI: number analyzed (Participants) | 0 | 3 | 0 | 3
    SAVI |  | 0.786 (0.275) |  | 0.786 (0.275)
    AGS: number analyzed (Participants) | 0 | 0 | 2 | 2
    AGS |  |  | 0.705 (0.77) | 0.705 (0.77)
Pre- Treatment Period:Baseline (Average) Mean Daily Diary Score [Mean (Standard Deviation); unit: score on a scale] — For CANDLE, participant or caregiver was instructed to rate each symptom (fever, rash, musculoskeletal pain, headache and fatigue in the diary on a scale from 0 to 4 (where a score of 0 = no symptoms, 1 = mild symptoms, 2 = moderate symptoms, 3 = more severe symptoms, and 4 = severe symptoms [equivalent to "worst" symptoms]. The mean daily score range was 0-4 with the higher score indicating a more severe symptom. Total score was not utilized. Population: SAVI and AGS did not have Pre-treatment period data therefore only CANDLE cohort data were collected.
  score on a scale
    number analyzed (Participants) | 5 | 0 | 0 | 5
    (all) | 0.642 (0.322) |  |  | 0.642 (0.322)
Pre-Treatment Period:Baseline (Average) Physician's Global Assessment of Disease Activity Scores [Mean (Standard Deviation); unit: score on a scale] — The Physician's Global Assessment of Disease Activity is used to assess the patient's current disease activity, as it relates to their signs and symptoms. The instrument uses a 21-circle Visual Analog Scale (VAS) ranging from 0 to 10 (using 0.5 increments) where 0 = "no activity" and 10 = "maximum activity" (Filocamo et al. 2010). Higher scores indicate greater disease severity. Population: SAVI and AGS did not have Pre-treatment period data therefore only CANDLE cohort data were collected.
  score on a scale
    number analyzed (Participants) | 5 | 0 | 0 | 5
    (all) | 5.45 (1.33) |  |  | 5.45 (1.33)
Pre-Treatment Period: Baseline (Average) % of days where participants' daily diary score was < 0.5. [Mean (Standard Deviation); unit: Percentage (%) of days] — Baseline (Average) Percentage of Days Meeting the Criteria of Participant's Mean Daily Diary Score <0.5 was reported. Population: SAVI and AGS did not have Pre-treatment period data therefore only CANDLE cohort data were collected.
  Percentage (%) of days
    number analyzed (Participants) | 5 | 0 | 0 | 5
    (all) | 35.6 (24.4) |  |  | 35.6 (24.4)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Daily Diary Scores in Participants With CANDLE (Primary Treatment Period)
Description: Diaries were specific to individual indications or conditions (i.e., NNS/CANDLE, SAVI, or AGS). For NNS/CANDLE, participant or caregiver was instructed to rate each symptom (fever, rash, musculoskeletal pain, headache and fatigue in the diary on a scale from 0 to 4 (where a score of 0 = no symptoms, 1 = mild symptoms, 2 = moderate symptoms, 3 = more severe symptoms, and 4 = severe symptoms [equivalent to "worst" symptoms]. The mean daily score range was 0-4 with the higher score indicating a more severe symptom. Total score was not utilized.
Time Frame: Baseline, 20 weeks
Population: CANDLE: All enrolled participants who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CANDLE
Number analyzed (Participants) | 5
score on a scale | -0.217 (0.586)

2. Primary Outcome: Change From Baseline in Mean Daily Diary Scores in Participants With SAVI (Primary Treatment Period)
Description: Diaries were specific to individual indications or conditions (i.e. NNS/CANDLE, SAVI, or AGS). For SAVI, participant or caregiver was instructed to rate each symptom (fever, rash, musculoskeletal pain, fatigue, respiratory/breathing problems, and ulcers/ischemic lesions in the diary on a scale from 0 to 4 (where a score of 0 = no symptoms, 1 = mild symptoms, 2 = moderate symptoms,3 = more severe symptoms, and 4 = severe symptoms [equivalent to "worst" symptoms].The mean daily score range was 0-4 with the higher score indicating a more severe symptom. Total score was not utilized.
Time Frame: Baseline, 32 weeks
Population: SAVI: All enrolled participants who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SAVI
Number analyzed (Participants) | 3
score on a scale | -0.23 (0.238)

3. Primary Outcome: Change From Baseline in Mean Daily Diary Scores in Participants With AGS (Primary Treatment Period)
Description: Diaries were specific to individual indications or conditions (i.e. NNS/CANDLE, SAVI, or AGS). For AGS, participant or caregiver was instructed to rate each symptom (rating) (neurologic disability (0, 5, 7,10) crying (0, 1, 2, 3), length of uninterrupted sleep (0, 1, 2, 3), generalized seizure (0, 8), fever (0,1), excessive irritability (0, 1, 2, 3), skin findings(body) (0, 1, 2, 3), and skin findings (hands, feet, and ears) (0, 1, 2, 3) with a higher score for each symptom indicating a more severe symptom. The mean daily diary score was the average of all symptom scores and the range was 0 - 4.25 with the higher score indicating a more severe symptom. Total score was not utilized.
Time Frame: Baseline, 32 weeks
Population: AGS: All enrolled participants who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aicardi-Goutières Syndrome (AGS)
Number analyzed (Participants) | 2
score on a scale | -0.045 (0.164)

4. Secondary Outcome: Change From Baseline in Mean Daily Diary Scores in Participants With CANDLE (Primary Treatment and Maintenance Period)
Description: as for outcome 1
Time Frame: Baseline, 191.1 weeks
Population: CANDLE: All enrolled participants who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CANDLE
Number analyzed (Participants) | 5
score on a scale | -0.24 (0.613)

5. Secondary Outcome: Change From Baseline in Mean Daily Diary Scores in Participants With SAVI (Primary Treatment and Maintenance Period)
Description: as for outcome 2
Time Frame: Baseline, 202.9 weeks
Population: SAVI: All enrolled participants who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SAVI
Number analyzed (Participants) | 3
score on a scale | -0.286 (0.333)

6. Secondary Outcome: Change From Baseline in Mean Daily Diary Scores in Participants With AGS (Primary Treatment and Maintenance Period)
Description: as for outcome 3
Time Frame: Baseline, 206.1 weeks
Population: AGS: All enrolled participants who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aicardi-Goutières Syndrome (AGS)
Number analyzed (Participants) | 2
score on a scale | -0.08 (0.114)

7. Secondary Outcome: Number of Participants With Decrease in Daily Dose of Corticosteroids in Participants With CANDLE, SAVI and AGS (Primary Treatment Period)
Description: Decrease was defined as total steroid dose at the visit <0.15 mg/kg/day (prednisone-equivalent) or >=50% decrease from baseline.
Time Frame: CANDLE: Week 20, SAVI and AGS: Week 32
Population: CANDLE, SAVI and AGS: All enrolled participants who received at least one dose of study drug and took corticosteroids at baseline with evaluable data for this outcome.
Measure: Number; unit: participants
Arm/Group | CANDLE | SAVI | Aicardi-Goutières Syndrome (AGS)
Number analyzed (Participants) | 5 | 1 | 1
participants | 4 | 1 | 1

8. Secondary Outcome: Number of Participants With Decrease in Daily Dose of Corticosteroids in Participants With CANDLE, SAVI and AGS (Primary Treatment and Maintenance Period)
Description: Decrease was defined as total steroid dose <0.15 mg/kg/day (prednisone-equivalent) or >=50% decrease from baseline.
Time Frame: CANDLE: Week 191.1; SAVI: 202.9 and AGS: Week 206.1
Population: as for outcome 7
Measure: Number; unit: participants
Arm/Group | CANDLE | SAVI | Aicardi-Goutières Syndrome (AGS)
Number analyzed (Participants) | 5 | 1 | 1
participants | 3 | 1 | 1

9. Secondary Outcome: Change From Baseline in Patient's Symptom Specific Daily Diary Scores For Participants With CANDLE (Primary Treatment Period)
Description: Diaries were specific to individual indications or conditions (i.e, NNS/CANDLE,SAVI, or AGS). For NNS/CANDLE, participant or caregiver was instructed to rate each symptom (fatigue, fever, headache, musculoskeletal pain and rash in the diary on a scale from 0 to 4, where a score of 0 = no symptoms, 1 = mild symptoms, 2 = moderate symptoms, 3 = more severe symptoms, and 4 = severe symptoms [equivalent to "worst" symptoms]). The mean daily score range was 0-4 with the higher score indicating a more severe symptom.
Time Frame: Baseline, 20 weeks
Population: CANDLE: All enrolled participants who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CANDLE
Number analyzed (Participants) | 5
score on a scale
  Fatigue | -0.029 (0.997)
  Fever | 0 (0)
  Headache | 0.057 (0.128)
  Musculo-skeletal Pain | -0.514 (1.128)
  Rash | -0.6 (0.894)

10. Secondary Outcome: Change From Baseline in Patient's Symptom Specific Daily Diary Scores For Participants With SAVI (Primary Treatment Period)
Description: Diaries were specific to individual indications or conditions (i.e. NNS/CANDLE, SAVI, or AGS). For SAVI, participant or caregiver was instructed to rate each symptom (fatigue, fever, musculoskeletal pain, rash, respiratory/breathing problems, and ulcers/ischemic lesions in the diary on a scale from 0 to 4, where a score of 0 = no symptoms, 1 = mild symptoms, 2 = moderate symptoms, 3 = more severe symptoms, and 4 = severe symptoms [equivalent to "worst" symptoms]). The mean daily score range was 0-4 with the higher score indicating a more severe symptom.
Time Frame: Baseline, 32 weeks
Population: SAVI: All enrolled participants who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SAVI
Number analyzed (Participants) | 3
score on a scale
  Fatigue | -0.381 (0.541)
  Fever | -0.095 (0.165)
  Musculo-skeletal Pain | -0.238 (0.412)
  Rash | -0.333 (0.577)
  Respiratory / Breathing Symptoms | -0.333 (0.577)
  Ulcers / Ischemic Lesions | 0 (0)

11. Secondary Outcome: Change From Baseline in Patient's Symptom Specific Daily Diary Scores For Participants With AGS (Primary Treatment Period)
Description: Diaries were specific to individual indications or conditions (i.e. NNS/CANDLE, SAVI, or AGS). For AGS, participant or caregiver was instructed to rate each symptom (rating) (crying (0, 1, 2, 3), excessive irritability (0, 1, 2, 3), fever (0,1), generalized seizure (0, 8), length of uninterrupted sleep (0, 1, 2, 3), neurologic disability (0, 5, 7,10), skin findings(body) (0, 1, 2, 3), and skin findings (hands, feet, and ears) (0, 1, 2, 3) with a higher score for each symptom indicating a more severe symptom.
Time Frame: Baseline, 32 weeks
Population: AGS: All enrolled participants who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aicardi-Goutières Syndrome (AGS)
Number analyzed (Participants) | 2
score on a scale
  Crying | 0 (0)
  Excessive Irritability | 0 (0)
  Fever | -0.071 (0.101)
  Generalized Seizure | 0 (0)
  Length of Uninterrupted Sleep | 0.286 (0.404)
  Neurologic Disability | 0 (0)
  Skin Findings (Body) | -0.5 (0.707)
  Skin Findings (Hands, Feet, Ears) | -0.071 (0.101)

12. Secondary Outcome: Change From Baseline in Patient's Symptom Specific Daily Diary Scores For Participants With CANDLE (Primary Treatment and Maintenance Period)
Description: as for outcome 9
Time Frame: Baseline, 191.1 weeks
Population: CANDLE: All enrolled participants who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CANDLE
Number analyzed (Participants) | 5
score on a scale
  Fatigue | -0.057 (1.172)
  Fever | 0 (0)
  Headache | 0.057 (0.128)
  Musculo-skeletal Pain | -0.514 (1.128)
  Rash | -0.686 (0.842)

13. Secondary Outcome: Change From Baseline in Patient's Symptom Specific Daily Diary Scores For Participants With SAVI (Primary Treatment and Maintenance Period)
Description: as for outcome 10
Time Frame: Baseline, 202.9 weeks
Population: SAVI: All enrolled participants who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SAVI
Number analyzed (Participants) | 3
score on a scale
  Fatigue | -0.381 (0.541)
  Fever | -0.095 (0.165)
  Musculo-skeletal Pain | -0.238 (0.412)
  Rash | -0.333 (0.577)
  Respiratory / Breathing Symptoms | -0.667 (1.155)
  Ulcers / Ischemic Lesions | 0 (0)

14. Secondary Outcome: Change From Baseline in Patient's Symptom Specific Daily Diary Scores For Participants With AGS (Primary Treatment and Maintenance Period)
Description: as for outcome 11
Time Frame: Baseline, 206.1 weeks
Population: AGS: All enrolled participants who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aicardi-Goutières Syndrome (AGS)
Number analyzed (Participants) | 2
score on a scale
  Crying | 0 (0)
  Excessive Irritability | 0 (0)
  Fever | -0.071 (0.101)
  Generalized Seizure | 0 (0)
  Length of Uninterrupted Sleep | 0 (0)
  Neurologic Disability | 0 (0)
  Skin Findings (Body) | -0.5 (0.707)
  Skin Findings on (Hands, Feet, Ears) | -0.071 (0.101)

15. Secondary Outcome: Change From Baseline in the Physician's Global Assessment of Disease Activity Scores in Participants With CANDLE (Primary Treatment Period)
Description: The Physician's Global Assessment of Disease Activity is used to assess the patient's current disease activity, as it relates to their signs and symptoms. The instrument uses a 21-circle Visual Analog Scale (VAS) ranging from 0 to 10 (using 0.5 increments) where 0 = "no activity" and 10 = "maximum activity" (Filocamo et al. 2010). Higher scores indicate greater disease severity.
Time Frame: Baseline, 20 weeks
Population: CANDLE: All enrolled participants who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CANDLE
Number analyzed (Participants) | 5
score on a scale | -2.1 (0.82)

16. Secondary Outcome: Change From Baseline in the Physician's Global Assessment of Disease Activity Scores in Participants With SAVI and AGS (Primary Treatment Period)
Description: The Physician's Global Assessment of Disease Activity is used to assess the patient's current disease activity, as it relates to their signs and symptoms. The instrument uses a 21-circle VAS ranging from 0 to 10 (using 0.5 increments) where 0 = "no activity" and 10 = "maximum activity" (Filocamo et al. 2010). Higher scores indicate greater disease severity.
Time Frame: Baseline, 32 weeks
Population: SAVI and AGS: All enrolled participants who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SAVI | Aicardi-Goutières Syndrome (AGS)
Number analyzed (Participants) | 3 | 2
score on a scale | -1.33 (1.76) | -3 (3.54)

17. Secondary Outcome: Change From Baseline in the Physician's Global Assessment of Disease Activity Scores in Participants With CANDLE (Primary Treatment and Maintenance Period)
Description: as for outcome 15
Time Frame: Baseline, 191.1 weeks
Population: CANDLE: All enrolled participants who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CANDLE
Number analyzed (Participants) | 5
score on a scale | -2.6 (2.07)

18. Secondary Outcome: Change From Baseline in the Physician's Global Assessment of Disease Activity Scores in Participants With SAVI and AGS (Maintenance Period)
Description: as for outcome 16
Time Frame: SAVI: Baseline, 202.9 weeks; AGS: Baseline, 206.1 weeks
Population: SAVI and AGS: All enrolled participants who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SAVI | Aicardi-Goutières Syndrome (AGS)
Number analyzed (Participants) | 3 | 2
score on a scale | -1.5 (1.73) | -3.75 (3.89)

19. Secondary Outcome: Change of Percentage of Days Meeting the Criteria of Participant's Mean Daily Diary Score <0.5 Compared to That in Pre-treatment Period in Participants With CANDLE (Primary Treatment Period)
Description: Change of Percentage of Days Meeting the Criteria of Participant's Mean Daily Diary Score <0.5 Compared to that in Pre-treatment period in Participants with CANDLE was evaluated
Time Frame: Pre-treatment period (average of 12-week pre-treatment data), up to 20 weeks
Population: CANDLE: All enrolled participants who received at least one dose of study drug. SAVI and AGS did not have Pre-treatment period data therefore only CANDLE cohort data were collected.
Measure: Mean (Standard Deviation); unit: Percentage of Days
Arm/Group | CANDLE
Number analyzed (Participants) | 5
Percentage of Days | 4.4 (48.7)

20. Secondary Outcome: Change of Percentage of Days Meeting the Criteria of Participant's Mean Daily Diary Score <0.5 Compared to That in Pre-treatment Period in Participants With CANDLE (Primary Treatment and Maintenance Period)
Description: as for outcome 19
Time Frame: Pre-treatment period (average of 12-week pre-treatment data), up to 191.1 weeks
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Percentage of Days
Arm/Group | CANDLE
Number analyzed (Participants) | 5
Percentage of Days | 2.0 (47.1)

21. Secondary Outcome: Change From Baseline in Growth Velocity (Height and Weight Z Score) (Primary Treatment and Maintenance Period)
Description: The change from baseline in normalized scores for body weight or height is measured using Z-scores. A Z-score indicates how many standard deviations a person's height or body weight is above or below the average for their age and gender. Z-score which was calculated by (value - [mean of the population]) / [SD of the population] at a given age/sex.
  Interpretation:
  Z-score of 0: The measurement is equal to the population mean. Z-score less than 0: The measurement is below the population mean. Z-score greater than 0: The measurement is above the population mean. An increase in the Z-score for weight or height means that the weight or height of the participants has increased more than the standard population during the study. For study participants with Z-scores less than 0 at baseline, an increase in Z-score is considered a positive outcome. A Z-score within the range of -2 to +2 indicates that the height or weight is within the normal range.
Time Frame: CANDLE: Baseline, 191.1 weeks; SAVI: Baseline, 202.9 weeks and AGS: Baseline, 206.1 weeks
Population: CANDLE, SAVI and AGS: All enrolled participants who received at least one dose of study drug and had evaluable data for this outcome.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | CANDLE | SAVI | Aicardi-Goutières Syndrome (AGS)
Number analyzed (Participants) | 1 | 2 | 2
Z-score
  Height | 3.03 (NA) — Standard Deviation is not calculable as number of participants analyzed (n) =1 | 0.75 (0.88) | 0.13 (1.17)
  Weight | 0.92 (NA) — Standard Deviation is not calculable as n=1 | 1.17 (0.03) | 0.46 (1.16)

22. Secondary Outcome: Change From Pre-treatment Period in Mean Daily Diary Scores For Participants With CANDLE (Primary Treatment Period)
Description: Diaries were specific to individual indications or conditions (ie, NNS/CANDLE,SAVI, or AGS). For NNS/CANDLE, participant or caregiver was instructed to rate each symptom (fever, rash, musculoskeletal pain, headache and fatigue in the diary on a scale from 0 to 4 (where a score of 0 = no symptoms, 1 = mild symptoms, 2 = moderate symptoms, 3 = more severe symptoms, and 4 = severe symptoms [equivalent to "worst" symptoms]. The mean daily score range was 0-4 with the higher score indicating a more severe symptom.
Time Frame: Pre-treatment period (average of 12-week pre-treatment data), up to 20 weeks
Population: CANDLE: All participants who received at least one dose of study drug. SAVI and AGS did not have Pre-treatment period data therefore only CANDLE cohort data were collected.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CANDLE
Number analyzed (Participants) | 5
score on a scale | 0.061 (0.432)

23. Secondary Outcome: Change From Pre-treatment Period in Mean Daily Diary Scores For Participants With CANDLE (Primary Treatment and Maintenance Period)
Description: as for outcome 22
Time Frame: Pre-treatment period (average of 12-week pre-treatment data), up to 191.1 weeks
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CANDLE
Number analyzed (Participants) | 5
score on a scale | 0.038 (0.464)

24. Secondary Outcome: Change From Pre-treatment Period in the Physician's Global Assessment of Disease Activity Scores For Participants With CANDLE (Primary Treatment Period)
Description: as for outcome 15
Time Frame: Pre-treatment period (average of 12-week pre-treatment data), up to 20 weeks
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CANDLE
Number analyzed (Participants) | 5
score on a scale | -1.75 (0.83)

25. Secondary Outcome: Change From Pre-treatment Period in the Physician's Global Assessment of Disease Activity Scores For Participants With CANDLE (Primary Treatment and Maintenance Period)
Description: as for outcome 15
Time Frame: Pre-treatment period (average of 12-week pre-treatment data), up to 191.1 weeks
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CANDLE
Number analyzed (Participants) | 5
score on a scale | -2.25 (1.79)

ADVERSE EVENTS:
Time Frame: CANDLE: Baseline Up to 191.1 Weeks; SAVI: Baseline Up to 202.9 Weeks and AGS: Baseline Up to 206.1 Weeks
Description: All enrolled participants who received at least one dose of study drug. Based on the planned safety analysis, adverse events were collected per the treatment regimen, irrespective of dose. Gender specific events occurring only in male or female participants have had the number of participants at risk adjusted accordingly.
Arm/Group | CANDLE | SAVI | Aicardi-Goutières Syndrome (AGS)
All-Cause Mortality (participants affected / at risk) | 0/5 | 1/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 3/5 | 1/3 | 0/2
Other Adverse Events (participants affected / at risk) | 5/5 | 3/3 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CANDLE (N=5) | SAVI (N=3) | Aicardi-Goutières Syndrome (AGS) (N=2)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Atypical mycobacterial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bronchopulmonary aspergillosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | CANDLE (N=5) | SAVI (N=3) | Aicardi-Goutières Syndrome (AGS) (N=2)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (2)
Blepharitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis allergic (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 2 (3) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (2) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Xerosis (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Adenoviral conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bk virus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Covid-19 (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Cytomegalovirus chorioretinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (2) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Metapneumovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2) | 0 (0) | 2 (23)
Otitis media (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Parotitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Periodontitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Pneumonia cytomegaloviral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Tinea capitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tracheitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (17) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Bk polyomavirus test positive (Investigations) | 3 (3) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 2 (2) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (3) | 0 (0)
Lymphocyte count increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Weight increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Post herpetic neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Head banging (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Menstruation irregular (Reproductive system and breast disorders) | 1/1 (1) | 0 (0) | 0/1 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (2)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 2 (4) | 1 (1) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (4) | 0 (0) | 0 (0)
Rosacea (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Continuous haemodiafiltration (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Haematoma evacuation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Lung assist device therapy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Mechanical ventilation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Pneumonectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Tracheostomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was terminated early due to efficacy/effectiveness reasons.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2023-09-04): https://cdn.clinicaltrials.gov/large-docs/53/NCT04517253/Prot_002.pdf
  • Statistical Analysis Plan (2024-11-26): https://cdn.clinicaltrials.gov/large-docs/53/NCT04517253/SAP_003.pdf